CLINICAL TRIAL: NCT03004573
Title: Functioning of the Mirror Neurons System in Parkinson's Disease and Its Impact on the Social Cognition
Brief Title: Role of Deep Brain Stimulation on Social Cognition in Parkinsonian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69 HCL15_0760; 2016-A00143-48 (Other: ID-RCB)
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; emotional recognition; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental)
  Interventions: Other: Neuropsychological detailed tests with focus on social cognition

INTERVENTIONS:
Other: Neuropsychological detailed tests with focus on social cognition — MATTIS, MOCA, BREF, Light points test, PDQ39

SUMMARY:
Parkinson's disease (PD) is usually responsible of cognitive and behavioral non-motor signs with a major impact on the quality of life. Social cognition is a complex system relying on emotion recognition (neurons mirror system, NMS), the theory of mind (with its two parts: emotional and cognitive), but also on the social and cultural environment and the personal history. The first step in this model is represented by the NMS, which seems to be altered in PD patients for both positive and negative emotions as shown in our preliminary study. The investigator purpose is to investigate the role of the treatment (levodopa and deep brain stimulation) on the functioning of the NMS.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease with motor fluctuations and dyskinesias receiving deep-brain stimulation
* Social insurance

Exclusion Criteria:

* No affiliation to the social insurance
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
variation of the emotional recognition score (point lights test) before deep brain surgery | Baseline
variation of the emotional recognition score (point lights test) after deep brain surgery | 1 year

SECONDARY OUTCOMES:
PDQ39 score (Parkinson's Disease Questionnaire) | 1 year
  Quality of Life
MATTIS (dementia rating scale) score | 1 year
  Global cognition. The Clinical Dementia Rating or CDR is a numeric scale used to quantify the severity of symptoms of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Teodor Danaila, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Neurologie C Hôpital " Pierre Wertheimer ", Bron, France

IPD SHARING:
Plan to Share IPD: No